CLINICAL TRIAL: NCT05778708
Title: Tai-Chi and Aerobic Exercise to Improve Emotional Symptom Cluster in Late-stage Lung Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Chia-Chin Lin, Professor and Head, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UW22-583
Record Dates: First submitted 2023-02-11; First posted 2023-03-21 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Advanced Lung Non-Small Cell Carcinoma

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Except for the primary research assistant who will inform the patients of their group allocation, all researchers on the team will be blinded to patients' group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tai-Chi intervention group (Experimental): The standardized 16-form Yang-style Tai-Chi exercise set will be adopted.
  Interventions: Behavioral: Tai-Chi intervention
- Aerobic exercise intervention (Experimental): The aerobic exercise class will be designed to cover both aerobic and resistance exercises.
  Interventions: Behavioral: Aerobic exercise intervention
- Self-management control group (No Intervention): Patients in this group will receive written information regarding the recommended levels of exercise (i.e., at least 150 min of moderate-intensity or 75 min of vigorous-intensity aerobic exercise every week) that they can perform at home (self-management) while continuing to receive their standard treatment. They will also be provided with a daily exercise log to record their exercise type, frequency, and intensity.

INTERVENTIONS:
Behavioral: Tai-Chi intervention — The standardized 16-form Yang-style Tai-Chi exercise set will be adopted. Group classes will take place in a community center twice a week for 16 weeks, with each class lasting approximately 60 minutes. Classes will be taught by an experienced Tai-Chi master. Patients will be instructed to practice the Tai-Chi exercises at home at least 3 times a week (30 min each time for a total of 90 min). Patients will be provided with a daily exercise log to record their exercise type, frequency, and intensity.
  Arms: Tai-Chi intervention group
Behavioral: Aerobic exercise intervention — The aerobic exercise class will be designed to cover both aerobic and resistance exercises. Group classes will take place in an exercise center twice a week for 16 weeks, with each class lasting approximately 60 minutes. Each class will be led by a certified exercise specialist. Patients will be provided with a daily exercise log to record their exercise type, frequency, and intensity.
  Arms: Aerobic exercise intervention

SUMMARY:
The goal of this randomized controlled trial is to investigate the effects of Tai-Chi and aerobic exercise on the emotional symptom cluster, and the underlying mechanism of that cluster, in late-stage lung cancer patients. Participants will be randomized into one of three groups: 1) Tai-Chi group, 2) aerobic exercise group, or 3) self-management control group. Both the Tai-Chi and aerobic exercise groups will attend twice-weekly group classes for 16 weeks (32 total contact hours). The self-management control group will receive written information regarding the recommended level of physical activity.

DETAILED DESCRIPTION:
Late-stage lung cancer patients (n = 318) meeting the inclusion criteria will be recruited and randomized into one of three groups: 1) Tai-Chi group, 2) aerobic exercise group, or 3) self-management control group. Both the Tai-Chi and aerobic exercise groups will attend twice-weekly group classes for 16 weeks (32 total contact hours). The self-management control group will receive written information regarding the recommended level of physical activity. To evaluate the effectiveness of Tai-Chi and aerobic exercise in alleviating the emotional symptom cluster (primary outcome) and individual symptoms (sleep disturbance, anxiety, depression, fatigue), outcome measures will be conducted at baseline, 8 weeks (mid-point assessment), 16 weeks (post-intervention), and 28 weeks (12-weeks post-intervention). A linear mixed-effects model will be used to study the between-group differences in outcomes. In addition, emotion regulation, mindfulness, and cardiorespiratory fitness will be evaluated at each data collection point, and structural equation modeling will be used for subsequent mediation analysis to determine their mediating role in outcome changes. Qualitative interviews will be conducted to understand patients' experience and evaluation of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with stage IIIB or IV non-small cell lung cancer confirmed by pathology, with no other cancer diagnosis within the previous year;
* a current Eastern Cooperative Oncology Group Performance Status of 0-2;
* experience of sleep disturbance, anxiety, depression, and fatigue in the past week (rating of 1 or more on a 0-10 numeric rating scale [NRS] for each symptom);
* able to communicate in Cantonese, Mandarin, or English;
* conscious and alert

Exclusion Criteria:

* suffering from a condition that hinders exercise performance (e.g., active neurological disorder, recent heart attack);
* currently participating in any other exercise or mind-body classes; or 3) performing regular exercises, defined as at least 150 minutes of moderate-intensity exercise weekly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Emotional symptom cluster at 8 weeks | 8 weeks
  NRSs for assessing each symptom of sleep disturbance, anxiety, depression, and fatigue over the past 7 days will be used to measure emotional symptom cluster severity. Higher score indicates more severe symptoms.
Change from Baseline Emotional symptom cluster at 16 weeks | 16 weeks
  NRSs for assessing each symptom of sleep disturbance, anxiety, depression, and fatigue over the past 7 days will be used to measure emotional symptom cluster severity. Higher score indicates more severe symptoms.
Change from Baseline Emotional symptom cluster at 28 weeks | 28 weeks
  NRSs for assessing each symptom of sleep disturbance, anxiety, depression, and fatigue over the past 7 days will be used to measure emotional symptom cluster severity. Higher score indicates more severe symptoms.

SECONDARY OUTCOMES:
Change from Baseline Sleep disturbance at 8 weeks | 8 weeks
  Measured by the Pittsburg Sleep Quality Index. The total score ranges from 0-21, with higher scores denoting poorer sleep.
Change from Baseline Sleep disturbance at 16 weeks | 16 weeks
  Measured by the Pittsburg Sleep Quality Index. The total score ranges from 0-21, with higher scores denoting poorer sleep.
Change from Baseline Sleep disturbance at 28 weeks | 28 weeks
  Measured by the Pittsburg Sleep Quality Index. The total score ranges from 0-21, with higher scores denoting poorer sleep.
Change from Baseline Fatigue at 8 weeks | 8 weeks
  Measured by the Brief Fatigue Inventory. Higher score denotes worse fatigue level.
Change from Baseline Fatigue at 16 weeks | 16 weeks
  Measured by the Brief Fatigue Inventory. Higher score denotes worse fatigue level.
Change from Baseline Fatigue at 28 weeks | 28 weeks
  Measured by the Brief Fatigue Inventory. Higher score denotes worse fatigue level.
Change from Baseline Anxiety and depression at 8 weeks | 8 weeks
  Measured by the Hospital Anxiety and Depression Scale. Higher score denotes higher level of anxiety and depression.
Change from Baseline Anxiety and depression at 16 weeks | 16 weeks
  Measured by the Hospital Anxiety and Depression Scale. Higher score denotes higher level of anxiety and depression.
Change from Baseline Anxiety and depression at 28 weeks | 28 weeks
  Measured by the Hospital Anxiety and Depression Scale. Higher score denotes higher level of anxiety and depression.
Change from Baseline Emotion regulation at 8 weeks | 8 weeks
  Measured by the Emotion Regulation Questionnaire. Higher scores indicating greater usage of that strategy.
Change from Baseline Emotion regulation at 16 weeks | 16 weeks
  Measured by the Emotion Regulation Questionnaire. Higher scores indicating greater usage of that strategy.
Change from Baseline Emotion regulation at 28 weeks | 28 weeks
  Measured by the Emotion Regulation Questionnaire. Higher scores indicating greater usage of that strategy.
Change from Baseline Mindfulness at 8 weeks | 8 weeks
  Measured by the Five Facet Mindfulness Questionnaire-Short Form. Higher score denotes higher mindfulness experience.
Change from Baseline Mindfulness at 16 weeks | 16 weeks
  Measured by the Five Facet Mindfulness Questionnaire-Short Form. Higher score denotes higher mindfulness experience.
Change from Baseline Mindfulness at 28 weeks | 28 weeks
  Measured by the Five Facet Mindfulness Questionnaire-Short Form. Higher score denotes higher mindfulness experience.
Change from Baseline Cardiorespiratory fitness at 8 weeks | 8 weeks
  Measured by the six-minute walk test. The distance walked at the end of 6 minutes will be measured in meters.
Change from Baseline Cardiorespiratory fitness at 16 weeks | 16 weeks
  Measured by the six-minute walk test. The distance walked at the end of 6 minutes will be measured in meters.
Change from Baseline Cardiorespiratory fitness at 28 weeks | 28 weeks
  Measured by the six-minute walk test. The distance walked at the end of 6 minutes will be measured in meters.
Change from Baseline agility at 8 weeks | 8 weeks
  Measured by the timed up-and-go test; unit: second.
Change from Baseline agility at 16 weeks | 16 weeks
  Measured by the timed up-and-go test; unit: second.
Change from Baseline agility at 28 weeks | 28 weeks
  Measured by the timed up-and-go test; unit: second.
Change from Baseline strength at 8 weeks | 8 weeks
  Measured by the sit-to-stand test; unit: number of times.
Change from Baseline strength at 16 weeks | 16 weeks
  Measured by the sit-to-stand test; unit: number of times.
Change from Baseline strength at 28 weeks | 28 weeks
  Measured by the sit-to-stand test; unit: number of times.
Change from Baseline balance at 8 weeks | 8 weeks
  Measured by the single-leg standing test; ; unit: second.
Change from Baseline balance at 16 weeks | 16 weeks
  Measured by the single-leg standing test; ; unit: second.
Change from Baseline balance at 28 weeks | 28 weeks
  Measured by the single-leg standing test; ; unit: second.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Chin Lin, PhD,FAAN,RN, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No